CLINICAL TRIAL: NCT03670771
Title: Incidence and Prognostic Significance of Intraabdominal Pressure in Critically Ill Patients
Brief Title: Intraabdominal Pressure in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal sayed ahmed, doctor, Assiut University
Other Study IDs: critically ill patients
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Critical Illness; Intra-Abdominal Hypertension
MeSH Terms: conditions — Critical Illness; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Harrahill method for measuring of intraabdominal pressure — IAP obtained by using patient own urine as the transducing medium. One clamps the Foley catheter just above the urine collection bag. The tubing is then held at a position of 30-40 cm above the symphysis pubis and the clamp is released. The IAP is indicated by the height (in cm) of the urine column from the pubic bone. The meniscus should show respiratory variations.

SUMMARY:
This study is conducted to evaluate the incidence and prognostic significance of IAH in medical ICU patients.

DETAILED DESCRIPTION:
Increased Intra-abdominal pressure (IAP) is an important cause of morbidity and mortality in ICU patients with consequent pulmonary, hepatic, central nervous and renal system impairments.

The increase in IAP is rarely diagnosed in ICU and the lack of diagnosis of this condition may lead to the worsening of patient prognoses because of retardation of appropriate interventions .

The current literatures show conflicting cutoff values of IAP that predict AKI, possibly due to the fact that many studies were conducted before publishing of the first Consensus of IAH/ACS, which standardized the measurement method of IAP.

Intra-abdominal hypertension is defined as a sustained or repeated pathologic elevation of intra-abdominal pressure greater than 12 mmHg [Malbrain et al 2004, cheathamML et al 2007]. Intra-abdominal hypertension is graded as follows:

* Grade I Intra-abdominal pressure 12-15 mmHg.
* Grade II Intra-abdominal pressure 16-20 mmHg.
* Grade III Intra-abdominal pressure 21-25 mmHg.
* Grade IV Intra-abdominal pressure greater than 25 mmHg Various risk factors contribute to the development of IAH in medical ICU including; massive fluid resuscitation (> 3500 ml/24 h), ileus, respiratory, renal, or liver dysfunction, hypothermia, acidosis, anemia, oliguria, and hyperlactatemia .

ELIGIBILITY:
Inclusion Criteria:

• All patients admitted to the critical care unit of internal medicine department not listed in the exclusion criteria.

Exclusion Criteria:

* Patients diagnosed with ESRD on dialysis.
* Patients with contraindications for internal urethral catheterization as urethral injury.
* Patients who had an obvious increase in IAP as; pregnant women and obese with body mass index (BMI) > 32 kg/m2.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients admitted to ICU due to medical cause irrespective of age or sex will be included in the study with detailed history and compelete examination will be done ,ECG will be done
  , SPO2 and arterial lactate concentrations and blood gases will be recorded twice daily, intraabdominal pressure wil be measured every at ltime of admission and every 6 hours until discharge or death occured.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluate the incidence and prognostic significance of IAH in medical ICU patients. | one year
  occurance of death ,improvement or organ failure

REFERENCES:
- [Result] Ruiz Ferron F, Tejero Pedregosa A, Ruiz Garcia M, Ferrezuelo Mata A, Perez Valenzuela J, Quiros Barrera R, Rucabado Aguilar L. [Intraabdominal and thoracic pressure in critically ill patients with suspected intraabdominal hypertension]. Med Intensiva. 2011 Jun-Jul;35(5):274-9. doi: 10.1016/j.medin.2011.02.009. Epub 2011 Apr 15. Spanish. PMID 21497415